CLINICAL TRIAL: NCT01980888
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib in Combination With Bendamustine and Rituximab for Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Efficacy and Safety of Idelalisib in Combination With Bendamustine and Rituximab in Adults With Previously Untreated Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-312-0123; 2013-003313-17 (EudraCT Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Idelalisib+bendamustine+rituximab (Experimental): Participants will receive idelalisib for 96 weeks plus bendamustine+rituximab for 21 weeks.
  Interventions: Drug: Idelalisib; Drug: Bendamustine; Drug: Rituximab
- Placebo+bendamustine+rituximab (Placebo Comparator): Participants will receive placebo to match idelalisib for 96 weeks plus bendamustine+rituximab for 21 weeks.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Placebo

INTERVENTIONS:
Drug: Idelalisib — 150 mg tablet administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL-101
  Arms: Idelalisib+bendamustine+rituximab
Drug: Bendamustine — Administered intravenously at a starting dose of 90 mg/m^2 for up to 6 cycles. Dosing will be based on mg/m^2 of body surface area.
Drug: Rituximab — Single-use vials administered intravenously weekly starting at 375 mg/m^2 on Day 1 (Week 0) and 500 mg/m^2 thereafter for a total of 6 infusions
Drug: Placebo — Placebo to match idelalisib administered orally twice daily
  Arms: Placebo+bendamustine+rituximab

SUMMARY:
The primary objective of this study is to evaluate the progression-free survival in participants with previously untreated chronic lymphocytic leukemia (CLL) who would otherwise be suitable for bendamustine and rituximab treatment as standard of care.

An increased rate of deaths and serious adverse events (SAEs) among participants with front-line CLL and early-line indolent non-Hodgkin lymphoma (iNHL) treated with idelalisib in combination with standard therapies was observed by the independent data monitoring committee (DMC) during regular review of 3 Gilead Phase 3 studies. Gilead reviewed the unblinded data and terminated this study in agreement with the DMC recommendation and in consultation with the US Food and Drug Administration (FDA).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of B-cell CLL, with diagnosis established according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL)
* No prior therapy for CLL other than corticosteroids for disease complications
* CLL that warrants treatment
* Presence of measurable lymphadenopathy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Key Exclusion Criteria:

* Known histological transformation from CLL to an aggressive lymphoma (ie, Richter transformation)
* Known presence of myelodysplastic syndrome
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of randomization
* Ongoing liver injury
* History of non-infectious pneumonitis
* Ongoing inflammatory bowel disease
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy other than corticosteroids
* Received last dose of study drug on another therapeutic clinical trial within 30 days prior to randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (91):
- United States (23):
  - St. Jude Heritage Healthcare Virginia K. Crosson Cancer Center, Fullerton, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Georgetown University, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Florida Cancer Specialists-South, Sarasota, Florida
  - Franciscan Physician Network Oncology & Hematology, Indianapolis, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hematology /Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Sarah Cannon Research Institute, Cincinnati, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Saint Francis Hospital, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (9):
  - St Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - Jarrett Street Specialist Centre, North Gosford, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Haematology and Bone Marrow Transplant Unit, Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Department of Haematology, Level 6, Bedford Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Frankston Hospital, Frankston, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
- Belgium (3):
  - Z N A Stuivenberg, Antwerp
  - AZ Sint-Jan AV Brugge-Oostende, Bruges
  - University Hospital Leuven, Leuven
- Canada (5):
  - Cancercare Manitoba - Maccharles Unit, Winnipeg, Manitoba
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - CHU de Québec - Hôpital de l'Enfant-Jésus, Québec, Quebec
- Croatia (3):
  - Klinicka bolnica Dubrava, Zagreb
  - Klinicka bolnica Merkur, Zagreb
  - UHC Zagreb, Zagreb
- Czechia (5):
  - Faculty hospital Ostrava, Ostrava-Poruba, Moravian-Silesian
  - University Hospital, Brno
  - Faculty Hospital Hradec Kralove, Hradec Králové
  - Faculty Hospital Plzen, Pilsen
  - Faculty Hospital Kralovske Vinohrady, Prague
- France (3):
  - CHRU de Lille, Hopital Claude Huriez, Lille
  - Hospital Saint-Louis, Paris
  - CHU Bretonneau, Tours
- Hungary (8):
  - Szent Borbála Hospital, Tatabánya, Komárom-Esztergom
  - Kaposi Mor Oktato Korhaz, Intezeti Gyogyszertar,, Kaposvár, Somogy County
  - Semmelweis University, Budapest
  - National Institute of Oncology, Budapest
  - University of Debrecen HSC Institute of internal Medicine, Department of Hematology, Debrecen
  - Pandy Kalman Hospital, Gyula
  - University Of Pecs, Medical School, Pécs
  - Szegedi Tudomanyegyetem AOK - Szent-Gyorgyi Albert Klinikai Kozpont, II. Belgyógyászati Klinika, Szeged
- Italy (5):
  - IRCCS Istituto Tumori, Bari, Apulia
  - Ospedale Oncologico Armando Businco, Cagliari
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - AOU Maggiore della Carità, Novara
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika Klinika Hematologii, Lodz
  - Centralny Szpital Kliniczny MSW w Warszawie Klinika Onkologii i Hematologii, Warsaw
  - Centrum Onkologii-Instytut Marii Sklodowskiej -Curie klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu Klinika i Katedra Hematologii,Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
  - Dolnoslakie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- Romania (2):
  - Emergency County Clinical Hospital Brasov, Brasov
  - Spitalul Clinic Colentina, Bucharest
- Spain (9):
  - Hospital Vall de Hebron, Barcelona, Catalonia
  - Hospital Clinic, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO, Hospitalet de Llobregat, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Puerta De Hierro, Madrid
- United Kingdom (9):
  - University College London, London, England
  - East Kent Hospitals University NHS Foundation Trust, Canterbury, Kent
  - Royal Marsden NHS Trust, Sutton, Surrey
  - University Hospital of Wales, Cardiff
  - Royal Liverpool & Broadgreen Univ. Hospitals NHS Trust, Liverpool
  - Hammersmith Hospitals NHS Trust, London
  - Oxford University Hospitals, Oxford
  - University Hospital Southampton NHS Trust, Southampton
  - Royal Wolverhampton Hospital NHS Trust, New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the North America, Australia, and Europe. The first participant was screened on 05 February 2014. The last study visit occurred on 16 June 2016.
Pre-assignment Details: 392 participants were screened.
Groups:
- Idelalisib+Bendamustine+Rituximab: Idelalisib (Zydelig®) 150 mg tablet twice daily + bendamustine intravenously (starting dose of 90 mg/m^2 for up to 6 total cycles) + rituximab (375 mg/m^2 on Day 1 and 500 mg/m^2 thereafter for at total of 6 infusions)
- Placebo+Bendamustine+Rituximab: Placebo tablet twice daily + bendamustine intravenously (starting dose of 90 mg/m^2 for up to 6 total cycles) + rituximab intravenously (375 mg/m^2 on Day 1 and 500 mg/m^2 thereafter for at total of 6 infusions)
Period: Overall Study
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Started | 157 | 154
Completed | 13 (Completed = reached primary efficacy endpoint of progressive disease or death.) | 21 (Completed = reached primary efficacy endpoint of progressive disease or death.)
Not Completed | 144 | 133
Not completed — Study Terminated by Sponsor | 116 | 122
Not completed — Withdrew Consent | 17 | 6
Not completed — Investigator's Discretion | 8 | 3
Not completed — Non-Compliance with Study Drug | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set: who were randomized regardless of whether subjects received any study drug(s), or received a different regimen from the regimen to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab | Total
Number analyzed (Participants) | 157 | 154 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.7) | 63 (10.0) | 64 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 48 | 105
  Male | 100 | 106 | 206
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 152 | 150 | 302
  Other | 3 | 1 | 4
  Not Permitted | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 2 | 13
  Not Hispanic or Latino | 146 | 149 | 295
  Not Permitted | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Romania | 4 | 1 | 5
  Hungary | 24 | 21 | 45
  United States | 35 | 25 | 60
  United Kingdom | 7 | 13 | 20
  Spain | 19 | 15 | 34
  Canada | 11 | 8 | 19
  Czech Republic | 10 | 17 | 27
  Belgium | 3 | 3 | 6
  Poland | 15 | 18 | 33
  Italy | 5 | 3 | 8
  Australia | 15 | 19 | 34
  France | 4 | 5 | 9
  Croatia | 5 | 6 | 11
Rai Stage at Screening [Count of Participants; unit: Participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL) with higher stages reflecting increasing severity.
  Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis with lymphadenopathy, Rai Stage II: Lymphocytosis with hepatomegaly or splenomegaly, Rai Stage III: Lymphocytosis with anemia, Rai Stage IV: Lymphocytosis with thrombocytopenia.
  Participants
    Stage I | 28 | 30 | 58
    Stage II | 66 | 58 | 124
    Stage III | 25 | 32 | 57
    Stage IV | 38 | 34 | 72
IgHV Mutation [Count of Participants; unit: Participants] — The mutation status of the unique immunoglobulin gene (IgHV) rearrangement in the monoclonal proliferation of B-cells in CLL can be used to predict aggressiveness of the disease. Participants with a mutated IgHV gene usually have a less aggressive and more indolent disease, with longer overall survival. Participants with an unmutated IgHV gene usually have a more aggressive disease and shorter overall survival.
  Participants
    Mutated | 54 | 54 | 108
    Unmutated | 102 | 100 | 202
    Missing | 1 | 0 | 1
17p Deletion in CLL Cells [Count of Participants; unit: Participants] — Participants with CLL who have a 17p deletion lack a portion of the chromosome that acts to suppress cancer growth and is a recognized negative prognostic risk factor.
  Participants
    Absent | 146 | 145 | 291
    Present | 10 | 9 | 19
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the interval from randomization to the first documentation of definitive disease progression or death from any cause. Definitive disease progression is CLL progression based on standard criteria, excluding lymphocytosis alone. PFS was to be assessed by an independent review committee (IRC).
Time Frame: Up to 22 months
Population: Intent to Treat (ITT) analysis set: all participants who are randomized in the study with treatment group designated according to initial randomization.
  Due to early study termination, the prespecified efficacy analyses were not conducted. The PFS data presented are investigator assessments rather than IRC assessments.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Number analyzed (Participants) | 157 | 154
months | NA [19.3 to NA] — NA: not reached | NA [19.6 to NA] — NA: not reached

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the proportion of participants who achieve a confirmed complete or partial response. ORR was to be assessed by an IRC.
Time Frame: Up to 22 months
Population: The study was terminated in agreement with the FDA due to urgent safety measures. Complete data were not collected for any participant.
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Nodal Response Rate
Description: Nodal response rate is defined as the proportion of participants who achieve a 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters of index lesions. Nodal response rate was to be assessed by an IRC.
Time Frame: Up to 22 months
Population: as for outcome 2
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Complete Response Rate
Description: Complete response rate is defined as the proportion of participants who achieve a confirmed complete response. Complete response rate was to be assessed by an IRC.
Time Frame: Up to 22 months
Population: as for outcome 2
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval from randomization to death from any cause. Overall survival was to be assessed by an IRC.
Time Frame: Up to 22 months
Population: as for outcome 2
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Minimal Residual Disease Negativity Rate at Week 36
Description: Minimal residual disease (MRD) negativity rate is defined as the proportion of participants with MRD < 10^-4 assessed by flow cytometry in bone marrow at Week 36 after therapy initiation or at least 12 weeks after the last dose of rituximab or bendamustine (whichever is later) for participants receiving the final dose of rituximab after the original scheduled date. MRD negativity rate was to be assessed by an IRC.
Time Frame: Up to 22 months
Population: as for outcome 2
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 22 months plus 30 days
Description: Safety Analysis Set: participants who received at least 1 dose of study treatment, with treatment assignments designated according to the actual treatment received.
Arm/Group | Idelalisib+Bendamustine+Rituximab | Placebo+Bendamustine+Rituximab
Serious Adverse Events (participants affected / at risk) | 113/156 | 68/154
Other Adverse Events (participants affected / at risk) | 154/156 | 150/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib+Bendamustine+Rituximab (N=156) | Placebo+Bendamustine+Rituximab (N=154)
Anaemia (Blood and lymphatic system disorders) | 8 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 29 | 16
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 3
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 26 | 19
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Unevaluable event (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 3
Hypersensitivity (Immune system disorders) | 0 | 1
Serum sickness (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Cytomegalovirus gastritis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Myocarditis infectious (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 5 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 6
Pneumonia fungal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 9 | 2
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Strongyloidiasis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
General physical condition abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 5 | 4
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Procedural pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Aortitis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib+Bendamustine+Rituximab (N=156) | Placebo+Bendamustine+Rituximab (N=154)
Anaemia (Blood and lymphatic system disorders) | 40 | 29
Neutropenia (Blood and lymphatic system disorders) | 84 | 90
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 16
Atrial fibrillation (Cardiac disorders) | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 14
Constipation (Gastrointestinal disorders) | 26 | 34
Diarrhoea (Gastrointestinal disorders) | 63 | 46
Dry mouth (Gastrointestinal disorders) | 11 | 4
Dyspepsia (Gastrointestinal disorders) | 15 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 4
Nausea (Gastrointestinal disorders) | 61 | 63
Stomatitis (Gastrointestinal disorders) | 10 | 4
Vomiting (Gastrointestinal disorders) | 37 | 23
Asthenia (General disorders) | 21 | 9
Chills (General disorders) | 21 | 14
Fatigue (General disorders) | 43 | 44
Mucosal inflammation (General disorders) | 14 | 1
Oedema peripheral (General disorders) | 19 | 16
Pyrexia (General disorders) | 71 | 38
Drug hypersensitivity (Immune system disorders) | 8 | 2
Bronchitis (Infections and infestations) | 5 | 8
Influenza (Infections and infestations) | 6 | 8
Nasopharyngitis (Infections and infestations) | 8 | 14
Oral candidiasis (Infections and infestations) | 8 | 4
Oral herpes (Infections and infestations) | 5 | 8
Pneumonia (Infections and infestations) | 10 | 3
Respiratory tract infection (Infections and infestations) | 9 | 4
Sinusitis (Infections and infestations) | 9 | 4
Upper respiratory tract infection (Infections and infestations) | 25 | 21
Urinary tract infection (Infections and infestations) | 15 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 21 | 33
Alanine aminotransferase increased (Investigations) | 22 | 3
Aspartate aminotransferase increased (Investigations) | 18 | 2
Neutrophil count decreased (Investigations) | 8 | 2
Weight decreased (Investigations) | 19 | 4
Decreased appetite (Metabolism and nutrition disorders) | 26 | 21
Dehydration (Metabolism and nutrition disorders) | 12 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 18
Dizziness (Nervous system disorders) | 13 | 13
Dysgeusia (Nervous system disorders) | 10 | 11
Headache (Nervous system disorders) | 16 | 25
Anxiety (Psychiatric disorders) | 11 | 9
Depression (Psychiatric disorders) | 8 | 2
Insomnia (Psychiatric disorders) | 17 | 12
Dysuria (Renal and urinary disorders) | 9 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 4
Erythema (Skin and subcutaneous tissue disorders) | 12 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 32
Rash (Skin and subcutaneous tissue disorders) | 63 | 34
Rash macular (Skin and subcutaneous tissue disorders) | 8 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 | 12
Hypotension (Vascular disorders) | 11 | 10

LIMITATIONS AND CAVEATS:
The study was terminated in agreement with the FDA due to urgent safety measures. Due to early study termination, the prespecified efficacy analyses were not conducted. The PFS data presented are investigator assessments rather than IRC assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years